CLINICAL TRIAL: NCT05113589
Title: Circadian Variation of Blood Pressure in Patients With Fibromyalgia After a Whole Body Photobiomodulation Treatment: a Triple-blinded Randomized Clinical Trial
Brief Title: Fibromyalgia and Circadian Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, SANTIAGO NAVARRO LEDESMA, UNIVERSITY PROFESSOR, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMCBP
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Blood Pressure
Keywords: blood pressure; autonomic symptoms; pain; fibromyalgia
MeSH Terms: conditions — Pain; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBM TREATMENT (Experimental): REAL PBM TREATMENT
  Interventions: Device: PBM TREATMENT
- PLACEBO PBM (Placebo Comparator): PLACEBO PBM TREATMENT
  Interventions: Device: PLACEBO PBM

INTERVENTIONS:
Device: PBM TREATMENT — Participants randomized to this treatment will receive a whole body PBM treatment using a NovoTHOR® whole body light bed. For each treatment session, participants will lie supine in the treatment bed for 20 minutes, with no or minimal attire (underwear). Treatment sessions will be three times weekly for a period of 4 weeks, totalling 12 treatment sessions
  Arms: PBM TREATMENT
Device: PLACEBO PBM — The placebo feature of the whole body PBM bed provides controls that select active or placebo (sham) treatments in a way undetectable by participant, operator or observers, such that no-one is aware whether the participant is receiving an active or placebo treatment. There is a switch box that randomises participants to active or placebo; no other randomisation is necessary.
  Arms: PLACEBO PBM

SUMMARY:
Fibromyalgia syndrome (FMS) is a chronic and multicomponent illness with unknown etiology and is considered the most frequent cause of diffuse chronic musculoskeletal pain. There is little evidence to confirm if the condition is fully improved after a specific treatment program. Thus a multifactorial understanding of the pathology is crucial to propose new alternative treatments. In this regard, an alteration in circadian blood pressure and persistent nocturnal sympathetic hyperactivity have been shown in patients suffering from fibromyalgia syndrome, leading to malfunctioning in the autonomic nervous system. This is a common pathogenesis shared also by patients with non-dipping blood pressure pattern, which has been closely associated with cardiovascular morbidity. Finally, a significant relationship between fibromyalgia syndrome and non-dipping blood pressure pattern has been shown. Therefore, alterations in circadian blood pressure appear as an additional risk factor in patients with fibromyalgia syndrome, and treatments focus on recovering such blood pressure pattern may be indicated.

DETAILED DESCRIPTION:
Studying variations of blood pressure is a way of assessing the master circadian clock, through the diurnal/nocturnal BP ratio.

When alteration of the circadian rhythm appears, neurohumoral factors that affect autonomic nervous and cardiovascular systems are affected, which presents persistent changes in the blood pressure pattern. These alterations caused by a disturbed circadian rhythm could contribute to the pathogenesis of chronic disorders in general and especially to fibromyalgia syndrome.

The aim of the study is to analyze changes in blood pressure and central sensitisation (pain pressure threshold) after a whole-body photobiomodulation treatment in patients suffering from fibromyalgia syndrome, as well as in pain, quality of life and autonomic symptoms. Furthermore, to study the level of association between blood pressure changes and pain perception, quality of life and autonomic symptoms after the end of the treatment. Finally, to study the effects of the treatment 3 months after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed from FM presenting generalized pain in at least four or five regions.
* Present symptoms for at least 3 months at similar levels.

Exclusion Criteria:

* Inflammatory, neurological, or orthopedic disease which can alter balance, hearing, and vision, and cognitive impairment in terms of the ability to answer questions.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change of Diurnal/nocturnal blood pressure ratio perceived at three months | time (t) 1(prior to treatment), t2 (immediately after treatment ), t3 (3 months after completion of treatment)
  The diurnal/nocturnal blood pressure ratio is defined as the nocturnal decline in BP relative to the diurnal blood pressure mean, and it is calculated as 100×(mean diurnal blood pressure-mean nocturnal blood pressure)/mean diurnal blood pressure. Mean blood pressure is calculated by mean blood pressure = diastolic pressure + 1/3 (systolic pressure - diastolic pressure).
  There are four possible groups: extreme-dippers (diurnal/nocturnal BP ratio ≥20%), normal dippers (ratio ≥10%), non-dippers (ratio <10%), and inverse-dippers or risers (ratio <0%, indicating nocturnal BP above the diurnal mean).

SECONDARY OUTCOMES:
Change from baseline perceived pain at 3 months | time (t) 1(prior to treatment), t2 (immediately after treatment ), t3 (3 months after completion of treatment)
  Visual Analogue Scale (VAS) is used by the patient to quantify the pain from 0 (without any pain) to 10 (the worst pain)
Change from autonomic nervous system activity at 3 months | time (t) 1(prior to treatment), t2 (immediately after treatment ), t3 (3 months after completion of treatment)
  The Autonomic Symptom Profile (ASP) is a validated self-report questionnaire that comprehensively assesses autonomic symptoms across 11 subscales and yields a composite autonomic symptom score, where higher scores mean a better outcome and lower scores mean a worst outcome. Autonomic nervous system activity provides quantitative information regarding cardiac autonomic tone.
Change from baseline Pain pressure threshold at 3 months | time (t) 1(prior to treatment), t2 (immediately after treatment ), t3 (3 months after completion of treatment)
  Tender points will be assessed using a standard pressure algometer (FPK 20; Wagner Instruments, Greenwich, CT, USA.): occiput at the suboccipital muscle insertions, low cervical at the anterior aspects of the intertransverse spaces at C5-C7, trapezius at the midpoint of the upper border, supraspinatus at origins, above the scapula spine near the medial border, paraspinous 3 cm lateral to the midline at the level of the mid-scapula, second rib at the second costochondral junctions, just lateral to the junctions on the upper surfaces, lateral pectoral at the level of the fourth rib at the anterior axillary line, lateral epicondylee 2 cm distal to the epicondyles and medial epicondyle at the epicondyles.
Change from elastography at 3 months | time (t) 1(prior to treatment), t2 (immediately after treatment ), t3 (3 months after completion of treatment)
  Quantified elastography in tender points. Changes in the status of myofascial trigger-points can be demonstrated with an objective and reproducible USE measure

CONTACTS AND LOCATIONS:
Overall Officials: SANTIAGO NAVARRO-LEDESMA, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Ana González Muñon, Málaga, Spain